CLINICAL TRIAL: NCT03119740
Title: Clinical Value of Postoperative C-reactive Protein in the Detection of Complications After Open and Laparoscopic Appendectomy
Brief Title: Postoperative Complications After Appendectomy
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Principal Investigator, Klugsberger Bettina, MD, Ludwig Boltzmann Institute for Operative Laparoscopy
Other Study IDs: APPCO-017
Record Dates: First submitted 2017-04-11; First posted 2017-04-19 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- open appendectomy: Patients were selected retrospectively on the basis of the documented MEL code (medical service code) of open appendectomy (AE)
- laparoscopic appendectomy: Patients were selected retrospectively on the basis of the documented MEL code (medical service code) of open laparoscopic appendectomy (LSK AE)

SUMMARY:
The frequency of complications after appendectomy is about 9% . The predictive value of CRP as an indicator of postoperative complications has been addressed in a small number of studies. The aim of the present retrospective analysis was to determine whether postoperative CRP levels are a reliable predictor of postoperative complications.

DETAILED DESCRIPTION:
Background: Acute appendicitis is a common emergency in general surgery. The frequency of complications after appendectomy is about 9% [9]. The predictive value of CRP as an indicator of postoperative complications has been addressed in a small number of studies. The aim of the present retrospective analysis was to determine whether postoperative CRP levels are a reliable predictor of postoperative complications.

Methods: This retrospective single-center cohort study comprised 744 patients who had undergone open or laparoscopic appendectomy for clinically suspected appendicitis between 1 January 2011 and 31 December 2015 at the department of general and visceral surgery, Kepler University Hospital in Linz, Austria. Demographic data, the surgical technique, postoperative complications, histopathological findings, postoperative white blood counts, and C-reactive protein levels were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* clinically suspected appendicitis between 1 January 2011 and 31 December 2015

Exclusion Criteria:

* an elective appendectomy as part of an oncological or gynecological operation tumor was found intraoperatively and required ileocecal resection or right hemicolectomy

Ages: 18 Years to 96 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients who had undergone open or laparoscopic appendectomy because of clinically suspected appendicitis between 1 January 2011 and 31 December 2015 at the department of general and visceral surgery, Kepler University Hospital in Linz, Austria
Sampling Method: Non-Probability Sample
Enrollment: 744 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
superficial wound infection | 4 weeks postoperative
  superficial wound infection in open and laparoscopic appendectomy

SECONDARY OUTCOMES:
intraabdominal abscess | 4 weeks postoperative
  intraabdominal abscess in open and laparoscopic appendectomy
ileus | 4 weeks postoperative
  ileus in open and laparoscopic appendectomy

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Shamiyeh, MD, Study Director — Clinic for General and Visceral Surgery, Kepler University Clinic Linz
Locations (1):
- Clinic for General and Visceral Surgery, Kepler University Clinic Linz, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barkhausen S, Wullstein C, Gross E. [Laparoscopic versus conventional appendectomy--a comparison with reference to early postoperative complications]. Zentralbl Chir. 1998;123(7):858-62. German. PMID 9746989
- [Background] Izbicki JR, Knoefel WT, Wilker DK, Mandelkow HK, Muller K, Siebeck M, Schweiberer L. Accurate diagnosis of acute appendicitis: a retrospective and prospective analysis of 686 patients. Eur J Surg. 1992 Apr;158(4):227-31. PMID 1352137
- [Background] Kaya B, Sana B, Eris C, Karabulut K, Bat O, Kutanis R. The diagnostic value of D-dimer, procalcitonin and CRP in acute appendicitis. Int J Med Sci. 2012;9(10):909-15. doi: 10.7150/ijms.4733. Epub 2012 Nov 13. PMID 23236260